CLINICAL TRIAL: NCT02929758
Title: The Effect of Speed of Processing Training on Pedestrian Behavior in Patients With Parkinson's Disease and Healthy Older Adults
Brief Title: Speed of Processing Training in Patients With Parkinson's Disease and Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amy Amara, MD, Assistant Professor of Neurology, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: X150203003; 5P30AG022838 (NIH)
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Initial Training Group (Active Comparator): Healthy Controls will receive initial SOPT training and will be compared against controls in the delayed training group and the PD subjects in the initial training group
  Interventions: Behavioral: Speed of processing training (SOPT)
- Control Delayed Training Group (Active Comparator): Healthy Controls will receive delayed SOPT training and will be compared against controls in the initial training group and the PD subjects in the delayed training group
  Interventions: Behavioral: Speed of processing training (SOPT)
- PD Initial Training Group (Other): PD subjects will received initial SOPT training and will be compared against PD subjects in the delayed training group and the control subjects in the initial training group
  Interventions: Behavioral: Speed of processing training (SOPT)
- PD Delayed Training Group (Other): PD subjects will receive delayed SOPT training and will be compared against PD subjects in the initial training group and the control subjects in the delayed training group
  Interventions: Behavioral: Speed of processing training (SOPT)

INTERVENTIONS:
Behavioral: Speed of processing training (SOPT) — This is a game-like program designed based on the UFOV. It consists of five activities (Sweep Seeker, Bird Safari, Jewel Diver, Master Gardener, and Road Tour). The duration of training will be 3 months. Participants will be encouraged to train at least three-times weekly for 1-hour blocks and must complete at least 20 training sessions over the course of the three months.
  Other Names: InSight (registered trademark of Posit Science, Inc.)

SUMMARY:
The purpose of this prospective, within-subject randomized cross-over design study is to determine if a computer training program (Speed of Processing Training - SOPT) improves safe pedestrian behavior in patients with Parkinson's disease and in healthy older adults in a virtual reality pedestrian environment. Pedestrian injury poses significant risk to healthy older adults and patients with Parkinson's disease. Several age-related changes, including slowing of visual processing speed, increase risky pedestrian behavior. This study will determine if SOPT improves pedestrian behavior in patients with Parkinson's disease and healthy older adults and evaluate the persistence of the SOPT training effects.

DETAILED DESCRIPTION:
Pedestrian injury poses significant risk to healthy older adults and patients with Parkinson's disease. Several age-related changes, including slowing of visual processing speed, increase risky pedestrian behavior. Persons with Parkinson's disease (PD) are at even higher risk of pedestrian injury due to motor and non-motor symptoms. Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by motor symptoms including slowness, tremor, stiffness, and balance problems. Visual processing speed abnormalities, anxiety, and cognitive problems are common non-motor symptoms.

The Useful Field of View (UFOV®) test is a measure of visual processing speed. The UFOV® test is performed on a touch-screen computer that displays objects in the central and peripheral visual fields for brief durations. Successful performance on the test requires integration of visual sensory information and higher-order cognitive processing. Our own research has shown that the UFOV® test performance correlates with pedestrian behavior in PD patients.

Speed of Processing Training (SOPT) is a computer-based training that uses visual exercises to improve cognitive processing. The training involves identifying and localizing visual information quickly in increasingly demanding visual displays. SOPT has been demonstrated to improve performance on the UFOV test in healthy older adults and PD patients. It is hypothesized that SOPT training will improve pedestrian safety in healthy older adults and PD patients.

In the proposed study, we will use a within-subject, randomized, controlled, cross-over design to evaluate if a computer training program (Speed of Processing Training - SOPT) improves safe pedestrian behavior in patients with Parkinson's disease and in healthy older adults in a virtual reality pedestrian environment and if the effects of training persist long-term.

ELIGIBILITY:
Inclusion Criteria Parkinson's disease Subjects:

* Subjects with a clinical diagnosis of idiopathic Parkinson's disease based on the presence of bradykinesia and one or both of the following: rest tremor and/or rigidity
* On stable medications for at least 4 weeks prior to entering the study and expected to not need any medication changes for the duration of the study
* Age ≥50 at the time of entry into the study
* Age of onset of Parkinson's disease 45 - 85 years old
* Asymmetric onset of PD
* Progressive motor symptoms of PD
* Hoehn and Yahr stages 1-4
* Ability to walk up and down a single stair step
* Access to a computer with internet

Exclusion Criteria Parkinson's disease Subjects:

* Atypical features indicative of a Parkinson's Plus disorder (Progressive Supranuclear Palsy, Multiple Systems Atrophy, Corticobasal Degeneration) including cerebellar signs, supranuclear gaze palsy, apraxia, prominent autonomic failure, or other cortical signs.
* Neuroleptic treatment at time of onset of Parkinsonism
* Active treatment with a neuroleptic at time of study entry
* History of multiple strokes with stepwise progression of Parkinsonism
* History of multiple head injuries
* Inability to walk without assistance, including a cane, wheelchair, or walker
* Cognitive dysfunction that would prevent subject's ability to perform virtual reality simulation, speed of processing training, or complete questionnaire
* Blindness
* Any medical condition that, based on discretion of the PI, would prevent the subject's ability to participate in the study

Inclusion Criteria Control Subjects:

* Age ≥50 at the time of entry into the study
* On stable medications for at least 4 weeks prior to entering the study and expected to not need any medication changes for the duration of the study
* Ability to walk up and down a single stair step
* Access to a computer with internet

Exclusion criteria Control Subjects:

* Parkinson's disease or other neurodegenerative disorder
* Inability to walk without assistance, including a cane, wheelchair, or walker
* Cognitive dysfunction that would prevent subject's ability to perform virtual reality simulation, speed of processing training, or complete questionnaires
* Blindness
* Any medical condition that, based on the discretion of the PI, would prevent the subject's ability to participate in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Time to contact | 3 months
  Difference in time to contact between baseline and immediate post-training assessments in PD and healthy controls

SECONDARY OUTCOMES:
Useful Field of View (UFOV) | 3 months
  Difference in UFOV total score between baseline and immediate post-training assessments in PD and healthy controls
Executive function (MoCA, Trails, Stroop) | 3 months
  Difference in MoCA, Trails, and Stroop between baseline and immediate post-training assessments in PD and healthy controls
Vigilance | 3 months
  Differences in vigilance as measured by psychomotor vigilance task between baseline and immediate post-training assessments in PD and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Amy Amara, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States